CLINICAL TRIAL: NCT07148739
Title: Ensuring Access to Optimal Therapy in Cystic Fibrosis: The ENACT Study
Brief Title: Ensuring Access to Optimal Therapy in CF: The ENACT Study
Acronym: ENACT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jennifer Guimbellot, Principal Investigator - MD, Arkansas Children's Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENACT-NP; 1R01HL171034-01A1 (NIH)
Record Dates: First submitted 2025-05-02; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Cystic Fibrosis (CF)
Keywords: Cystic Fibrosis; CF; CFTR modulator; Pediatric CF patients; Elexacaftor; Tezacaftor; Ivacaftor
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; tezacaftor, ivacaftor drug combination

STUDY DESIGN:
Intervention Model Description: This is a pilot and feasibility study to assess the association of drug concentration with side effects, and to assess the feasibility of the use of therapeutic drug monitoring to adjust dosing in individuals with side effects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Other): Participants may be enrolled in an observational one-visit study for association of concentration with side effects. Participants may proceed to a single arm study if they have side effects to assess the feasibility of adjusting dose to maintain concentrations within an estimated effective range. Once within the range, dosing is no longer adjusted. Side effects will be evaluated as described in the protocol.
  Interventions: Drug: Elexacaftor / Ivacaftor / Tezacaftor; Other: therapeutic drug monitoring

INTERVENTIONS:
Drug: Elexacaftor / Ivacaftor / Tezacaftor — This study will examine different dosing strategies and outcomes for triple combination CFTR modulator therapy using the drug(s) elexacaftor, tezacaftor, and/or ivacaftor in patients with cystic fibrosis.
  Other Names: Triple Combination CFTR Modulator Therapy; ETI - Elexacaftor/Tezacaftor/Ivacaftor
Other: therapeutic drug monitoring — Participants who consent to the therapeutic drug monitoring study will have their dose adjusted to remain within estimated effective concentrations.

SUMMARY:
This clinical trial is examining the action and effects of several new drugs in the treatment of cystic fibrosis in children. In addition, several genetic factors are examined. The hope is that the ability to determine prior to treatment those individuals who will or will not respond to existing therapies will avoid needless risk of side effects and the high cost of a potentially ineffective treatment regimen. Understanding the way these drugs work in the body and the best way to study them is critical to expanding the use of these drugs to all patients with cystic fibrosis (CF).

DETAILED DESCRIPTION:
Understanding variation in genetic response to pharmacological treatments and personalized CFTR modulator response is crucial to the optimization of the use of these novel compounds; expansion to all patients who might benefit from them; and development of predictive biomarkers. In addition, the ability to determine prior to treatment those individuals who will or will not respond to existing therapies will avoid needless risk of side effects and the high cost of a potentially ineffective treatment regimen. Understanding the way these drugs work in the body and the best way to study them and the downstream effects is critical to expanding the use of these drugs to all patients with cystic fibrosis (CF).

ELIGIBILITY:
Inclusion Criteria:

* documentation of CF diagnosis per CFF diagnostic criteria and known CFTR genotype
* age 2 years and older
* ability to provide written informed consent and/or assent (by subject and/or legal guardian)
* on a stable dose of triple combination CFTR modulator therapy for at least two weeks prior to Visit 1
* clinically stable lung disease, defined as no documented acute decrease in FEV1 > 10%, OR use of additional antibiotics (intravenous [IV] or oral [PO]) within 4 weeks prior to screening

Exclusion Criteria:

* recent significant unintentional weight loss, as determined by the investigator, in the 4 weeks prior to screening
* pregnant or breastfeeding female
* history of alcohol or substance abuse in the 6 months prior to screening
* participation in a study involving an investigational intervention within 28 days (or 5 half-lives, whichever is longer) prior to screening
* in the opinion of the Investigator, medical or psychiatric illness, or other conditions that would interfere with participation

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Concentration (ng/mL) | One time assessment for observational part of the study, up to 6 times (6 months or more) for the therapeutic drug monitoring pilot and feasibility study.
  Drug concentration of CFTR modulators

SECONDARY OUTCOMES:
Participant Mental and Neuropsychological Health | From enrollment to the end of treatment at 6-12 months.
  Participants will respond to questionnaires about anxiety, depression, suicidal ideation and other indicators of mental and neuropsychological health. Participants will complete assessments and an exam at each study visit.
Investigators will evaluate the feasibility of reducing dose to manage Neuropsychological Side Effects (NPSE). | From enrollment to study conclusion at 6-12 months (after all visits are completed).
  The primary goal will be to assess feasibility to monitor clinical outcomes, patient receptiveness, collection of samples, and concentration interpretation. Assessment of feasibility will include the patient acceptance of dose reduction using an acceptability questionnaire, turnaround for quantitation results by timely return of result, and clinical appropriateness for dose reduction (by monitoring clinical response).
Response to dosing adjustments | From enrollment to study conclusion at 6-12 months, after all visits are completed.
  Outcome includes symptom assessment, spirometry, sweat chloride, weight, and TC quantitation at Visits 2-6. Investigators will monitor patients for 6 visits to assess CF and NP symptom stability under the supervision of the licensed clinical psychologist and TC concentration variability over time. At each visit investigators will re-assess dosing strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer S Guimbellot, Medical Degree and License, Principal Investigator — Arkansas Children's Hospital Research Institute
Locations (2):
- United States (2):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No